CLINICAL TRIAL: NCT03550599
Title: Adequacy of Pain Treatment in Radiotherapy: an Observational, Prospective, Multicenter Study (ARISE)
Brief Title: Adequacy of Pain Treatment in Radiotherapy
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Responsible Party: Principal Investigator, Alessio Giuseppe Morganti, Professor, IRCCS Azienda Ospedaliero-Universitaria di Bologna
Other Study IDs: ARISE
Record Dates: First submitted 2018-05-28; First posted 2018-06-08 (Actual); Last update posted 2019-01-14 (Actual); Status verified 2019-01

CONDITIONS: Cancer Pain; Analgesic Drugs
MeSH Terms: conditions — Cancer Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- patients accessing to Radiotherapy Unit: patients accessing to Radiotherapy Unit for oncologic treatment
  Interventions: Other: Patients accessing to Radiotherapy Unit

INTERVENTIONS:
Other: Patients accessing to Radiotherapy Unit — No intervention; information about patient and disease characteristics will be recorded as well as information about pain and analgesic treatment

SUMMARY:
Aim of the study is to evaluate adequacy of pain treatment in oncologic patients, accessing to Radiotherapy Unit

DETAILED DESCRIPTION:
Prescription of analgesic drugs is a basic topic in cancer patients, but undertreatment is common. The aim of the study is to analyse pain control and adequacy of antalgic treatments in patients coming to Radiotherapy Unit for radiation treatment.

ELIGIBILITY:
Inclusion Criteria:

- patients accessing to Radiotherapy Unit for radiation treatment (both palliative or with radical intent) with diagnosis of primitive or metastatic cancer;

Exclusion Criteria:

- Concomitant diseases that can affect reliability of collected data

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 2000 consecutive patients accessing to Radiotherapy Unit
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2018-03-01 (Actual); Primary Completion 2019-03-01 (Estimated); Study Completion 2019-06-01 (Estimated)

PRIMARY OUTCOMES:
Evaluation of adequacy of pain treatment | 2 months
  For all patients, Visual Analogue Scale (VAS) and information about type of analgesic drugs (no drugs; non-opioid drugs; weak opioids; strong opioids) will be recorded and analysed

CONTACTS AND LOCATIONS:
Overall Officials: Alessio G Morganti, MD, Principal Investigator — Radiation Oncology Center, Departement of Experimental, Diagnostic and Speciality Medicine-DIMES, University of Bologna, S.Orsola-Malpighi Hospital, Bologna, Italy
Locations (1):
- Radiation Oncology Center, Department of Experimental, Diagnostic and Speciality Medicine- DIMES, University of Bologna, S.Orsola-Malpighi Hospital, Bologna, BO, Italy

IPD SHARING:
Plan to Share IPD: No